CLINICAL TRIAL: NCT04907630
Title: The Effect of Antenatal Education Based on Improving Health Literacy on Adaptation of Pregnancy, General Self-Efficacy, Fear of Childbirth, and Health Literacy in Primiparous Pregnant Women: A Randomized Control Study
Brief Title: Antenatal Education Based on Improving Health Literacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Balikesir University (Other)
Responsible Party: Principal Investigator, Filiz Aslantekin Özçoban, Principal Investigator, Balikesir University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 0000-0002-040
Record Dates: First submitted 2021-05-22; First posted 2021-06-01 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Antenatal Education
Keywords: Health Literacy; Antenatal Education; General Self-Efficacy; Fear of Childbirth
MeSH Terms: interventions — Prenatal Education

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- intervention group-antenatal education of health literacy (HL-AE) (Experimental): It is the group that is given antenatal education based on improving health literacy (HL-AE).
  Interventions: Behavioral: Antenatal Education
- intervention group-Antenatal Education (AE) (Experimental): It is the group that gives antenatal education (AE)
  Interventions: Behavioral: Antenatal Education
- Control group (Experimental): No Intervention
  Interventions: Behavioral: Antenatal Education

INTERVENTIONS:
Behavioral: Antenatal Education — educational intervention
  Other Names: antenatal education based on improving health literacy

SUMMARY:
Aim: This study was aimed to evaluate the effect of antenatal education based on improving health literacy on the adaptation of pregnancy, general self-efficacy, fear of childbirth, and health literacy in primiparous pregnant women.

Design: It was a randomized controlled trial. Method: The research was carried out in a city located in the Marmara region of Turkey between July 2018 and April 2019. It was conducted with three groups, including one control (n=73) and two intervention groups (n=109). One of the intervention group was given antenatal education based on improving health literacy (n=53), and the other was only provided with antenatal education (n=56). Pregnancy Information Form, Prenatal Self-Evaluation Questionnaire, Pregnancy Related Anxiety Scale, General Self-Efficacy Scale, and Health Literacy-TR32 scale were used for data collection.

DETAILED DESCRIPTION:
Background: Pregnant women get themselves ready to give birth, maternity and parenting through antenatal education. These trainings make it easier to adapt to the processes in which pregnant women experience change. They also provide an important opportunity to support and maintain the competence and motivation to manage health responsibility.

Aim: To evaluate the impact of antenatal education intervention based on improving health literacy in order for primiparous pregnant women to; accept the pregnancy and adopt the role of maternity; increase the level of general self-efficacy and health literacy; reduce the fear of childbirth; and support the level of breastfeeding.

Design: It is an experimental and randomized controlled trial. Method: The research was carried out in a town located in the Marmara region of Turkey between April 2019 and July 2018. It was conducted with three groups, including one control (73) and two training groups (109). One of the training group was given antenatal education based on improving health literacy (HL-AE) (53), and the other was only provided with antenatal education (AE) (56). Pregnancy identification form, prenatal self-evaluation questionnaire, pregnancy related anxiety scale, general self-efficacy scale, Turkey health literacy -32 scale and postpartum data collection form were used for data collection.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer primiparous pregnant women
* 18 years and over,
* No have any disease
* In the second trimester

Exclusion Criteria:

* Not participating in five-week education,
* Any complications developed during the education period
* Voluntarily leaving.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Prenatal Self-Evaluation Questionnaire (PSEQ) | five weeks
  The scale was developed by Lederman et al. in 1979 to evaluate the adaptation of women to pregnancy and birth in the prenatal period (Lederman & Weis, 2009). The scale is a four-point Likert type consisting of seven subscales and 79 items. The highest score that can be obtained from the scale is 316 and the lowest one is 79. The Turkish validity and reliability of the scale was made by Beydağ and Mete (Cronbach's alpha=.83) (Beydağ & Mete, 2008).Two subscales of "acceptance of pregnancy" and "defining the role of maternity" were used for the research. Values that can be taken as an acceptance of pregnancy are between 14-56. Values that can be taken as the acceptance of the role of maternity are 15-60. A low score indicates that the mother's adaptation is better.
Fear of Childbirth and The Postpartum Period Scale | five weeks
  The scale was developed by Kitapçıoğlu et al in 2008 to evaluate the concerns about delivery and postpartum period. It is a five-point Likert-type scale. Scale includes 61 question items, and they are scored between 0-10 (Cronbach's alpha=.95). Decrease in the scale mean score shows that the concerns about childbirth are decreasing (Kitapçıoğlu et al., 2008).
General Self-Efficacy Scale | five weeks
  An original 23-item form was developed by Sherer et al (Sherer et al., 1982). The validity and reliability of the Turkish version was made by Yıldırım and İlhan, and a scale of 17 questions was created. The scale's total score ranges from 17 to 85 (Cronbach alpha=.80). The increase in the score shows that the belief in self-efficacy has increased (Yildirim & Ilhan, 2010).

SECONDARY OUTCOMES:
Turkey Health Literacy Scale-32 | five weeks
  It is a self-report scale developed to evaluate health literacy in adult individuals. The scale is based on the conceptual framework developed by the European Health Literacy Research Consortium. It was developed by Abacigil et al. (Cronbach alpha=.95). Each item is 4 degrees to indicate 1=Very easy, 2=Easy, 3=Hard, 4=Very hard. Codes were reversed when calculating the score. In terms of ease of calculation, the total score has been standardized with the help of the following formula to take a value between 0-50 (Abacigil et al., 2019).

CONTACTS AND LOCATIONS:
Locations (1):
- Balikesir University, Faculty of Health Sciences, Department of Midwifery Çağış Campus, Balıkesir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No